CLINICAL TRIAL: NCT03664401
Title: A Clinical Trial to Evaluate Kerecis Oral™ Compared to Autogenous Free Gingival Graft (AFGG) Tissue to Augment Gingival Soft Tissue and Wound Healing
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kerecis Ltd. (Industry)
Collaborators: Tufts University School of Dental Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 01-GING-001-Kerecis Oral
Record Dates: First submitted 2018-08-30; First posted 2018-09-10 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Mucogingival Deformity - Insufficient Keratinized Tissue

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled, split mouth (within subject) non-inferiority, single-center trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Kerecis Oral™ (Experimental): The Fish Skin Graft will be is cut to shape of wound bed and placed directly on the appropriate prepared recipient wound bed. The Fish skin graft has the smooth side down and the scaly side facing out. The graft will be sutured in place at either coronal end with resorbable sutures and may be secured apically if needed. A surgical dressing (Coe-Pak® ) will be placed over the graft if needed.
  Interventions: Device: Kerecis Oral™
- Autogenous Free Gingival Graft (Active Comparator): The recipient bed will be prepared at the appropriate sequential time as described. The graft will be harvested from the same side that the Free Gingival Graft is to be placed. A measurement will be made to determine the size of the donor tissue needed to be placed at the recipient site. Local anesthetic will be administered. The donor tissue will be harvested using the usual techniques. The width will be 5 mm and the length will match the predetermined measurement. The graft will be thinned as is usual practice.
  The harvested palatal graft will be centered on the study tooth and placed on the appropriately prepared recipient wound bed. The graft will be sutured with resorbable sutures on the mesial and distal aspects of the tooth. A surgical dressing (Coe-Pak® ) will be placed over the graft if needed.
  Interventions: Other: Free Gingival Graft

INTERVENTIONS:
Device: Kerecis Oral™
  Other Names: Acellular Fish Skin Graft
  Arms: Kerecis Oral™
Other: Free Gingival Graft — A free gingival autograft from patient palate placed and secured on wound bed
  Other Names: FGG
  Arms: Autogenous Free Gingival Graft

SUMMARY:
The purpose of this study is to evaluate Omega-3 Wound™ as an alternative to autogenous free gingival grafts harvested from the palate to treat human subjects with insufficient KT (< 2 mm)

DETAILED DESCRIPTION:
Primary objective:

The primary aim will be to see if Omega-3 Wound™ is clinically superior to tissue harvested from the palate (Autogenous Free Gingival Graft) when comparing before and after measurements of: keratinized tissue. Change in KT width from time of surgery to 6 months post-surgery (22).

Secondary objectives:

1. Measures of periodontal health (probing depth, recession levels, bleeding on probing, plaque score, clinical attachment level, resistance to muscle pull, vestibular depth, healing time) over 3 months (at study entry, 4 weeks, 3 months and 6 months)
2. Time of surgery
3. Subject Discomfort Survey during healing and at 1 week and 4 weeks
4. Subject Preference Questionnaire at month 6
5. Safety endpoints assessed by monitoring adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Age must be at least 18 years but no more than 70 years.
2. There must be at least two non-adjacent teeth in contralateral sides of the same jaw with an insufficient zone (≤ 2mm) of Keratinized gingiva that requires soft tissue grafting. (1-4 teeth may be treated). If adjacent teeth require grafting, only a single chosen tooth at each site will act as the test or control site, all teeth will however get the same treatment).
3. The goal of grafting will not be root coverage.
4. Females must have a documented negative urine pregnancy test if they are of childbearing potential.
5. All subjects must have read, understood and signed an Informed Consent Form (approved by the institutional review board (IRB)).
6. All subjects must be willing and able to follow study instructions and protocols.

Exclusion Criteria:

1. Any subject that has class III/IV recession with a shallow vestibule.
2. Any subject that has a vestibule depth of less than 7mm from the base of recession.
3. Any subjects with systemic conditions (i.e., diabetes mellitus, HIV, cancer, bone metabolic diseases) that typically precludes periodontal surgery.
4. Any subjects who are currently taking/received or have taken/received within two months prior to study entry, systemic corticosteroids, immunosupressive agents, radiation therapy, and/or chemotherapy which could compromise wound healing and preclude periodontal surgery. Any subjects taking intramuscular or intravenous bisphosphonates.
5. Any subjects with any acute lesions in the areas intended for surgery/or with a history of aphthous ulcers.
6. Any subjects who currently smoke.
7. Any subject with molar teeth that require treatment at the time of surgery.
8. Any subjects with teeth with Miller Grade =>2 mobility.
9. Any patients with known hypersensitivity to bovine collagen and/or iodine (shellfish allergy).
10. Any subjects who have received an investigational drug or biological/bioactive treatment within 30 days prior to study enrollment (medical or dental).
11. Any subjects previously treated with any allografts at the target site(s) or immediately adjacent teeth.
12. Any subjects who will not be able to complete the study per protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Change in KT width from time of surgery to 3 months post-surgery | 3 months
  Increase in KT Width in MM

SECONDARY OUTCOMES:
Probing depth | 3 months
  mm
Papillary height and widht | 3 months
  mm
Horizontal recession | 3 months
  mm
Subject completed discomfort questionaire | 3 months
  Standard questionare
Bleeding on probing | 3 months
  Y/N

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Karimbux, DMD, MMSc, Study Chair — Tufts University of Dental Medicine

IPD SHARING:
Plan to Share IPD: No